CLINICAL TRIAL: NCT03904667
Title: Application of Watson for Oncology in Hepatocellular Carcinoma Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20170101
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Liver Resection
Keywords: Watson artificial intelligence; hepatocellular carcinoma; surgical decisions
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Watson on oncology recommends surgery
  Interventions: Other: Watson on oncology surgery decision evaluation
- Watson on oncology does not recommend surgery
  Interventions: Other: Watson on oncology surgery decision evaluation

INTERVENTIONS:
Other: Watson on oncology surgery decision evaluation — Watson on oncology surgery decision evaluation. The system acquires and evaluates a large amount of structured and unstructured data from previous medical records through machine learning and natural language processing, and USES algorithms to select treatment options as the best choice for a particular patient.

SUMMARY:
The aim of this study was to evaluate the surgical decisions of Watson artificial intelligence in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatectomy is an effective treatment for patients with hepatocellular carcinoma, but liver failure after hepatectomy may lead to increased postoperative mortality. Therefore, it is very important to make preoperative surgical decisions, evaluate the safety of the operation and identify which patients are likely to suffer from liver failure. The artificial intelligence platform developed by IBM Watson for Watson tumor treatment decisions can provide treatment decisions and corresponding theoretical basis to guide surgical decisions based on the key clinical data of liver cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤ Age ≤80 years
2. Compling with the diagnosis criteria of complex hepatic carcinoma.
3. Primary hepatic carcinoma without intrahepatic or extrahepatic extensive cancer metastasis, the metastatic hepatic carcinoma whose primary focal has been controlled
4. Preoperative liver function is Child - Pugh grade A or B.
5. The patients are volunteered for the study.

Exclusion Criteria:

1. Patients with mental illness.
2. Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.)
3. The patients refused to take part in the study.
4. There are other co-existed malignant tumors.
5. Benign liver diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 hepatocellular carcinoma patients admitted to the department of hepatobiliary surgery of zhujiang hospital of southern medical university from January 2017 to December 2021 were selected and divided into experimental group and control group
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative outcomes | intraoperative
  Operative outcomes such as operative time, estimated blood loss and blood transfusion were recorded.

SECONDARY OUTCOMES:
Postoperative survival | 3 years
  Survival after hepatectomy

OTHER OUTCOMES:
Disease-free survival | 3 years
  Survival time without tumor after hepatectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China